CLINICAL TRIAL: NCT03721835
Title: A Multicenter, Post Market, Prospective Study Evaluating Safety and Efficacy of CONQUEST FN for the Treatment of Intracapsular Femoral Neck Fractures
Brief Title: Safety Study of Femoral Neck Fracture System
Acronym: CONQUEST FN
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow enrollment
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-3047-02
Record Dates: First submitted 2018-10-19; First posted 2018-10-26 (Actual); Results first posted 2023-09-25 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2021-02

CONDITIONS: Femoral Neck Fractures
Keywords: Femoral Neck Fracture; Hip; Broken hip; CONQUEST FN; Hip Fracture
MeSH Terms: conditions — Femoral Neck Fractures; Hip Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Control femoral neck fracture system (Other): This is a single arm study of subjects who are to be implanted with the CONQUEST FN™Femoral Neck Fracture System for treatment of a trauma related femoral neck fracture
  Interventions: Device: CONQUEST FN Femoral Neck Fracture System

INTERVENTIONS:
Device: CONQUEST FN Femoral Neck Fracture System — Fracture fixation device consisting of a single plate and three screws

SUMMARY:
The purpose of this study is to assess the reoperation rate of fractures that have occurred at the neck of the femur that are treated with the CONQUEST FN Femoral Neck Fracture System. The CONQUEST FN Femoral Neck Fracture System is approved for use by the United States Food and Drug Administration (FDA). It consists of a stainless steel plate and up to three (3) screws intended to treat both non-displaced and displaced fractures to the femoral neck.

DETAILED DESCRIPTION:
The CONQUEST FN™ represents the next generation femoral neck fracture system designed to offer better intra-operative reduction control with the assurance of eliminating device failure modes. This system is dedicated to treating both non-displaced and displaced intracapsular fractures of the femoral neck. It is a dynamic locked implant system that provides multiple points of fixed angle support with continuous compression across the fracture site, ensuring bone-on-bone contact during the fracture union process. The continuous fracture site compression and post-operative reduction maintenance is accomplished with the incorporation of telescoping compression screw technology. The novel system empowers surgeons to address the current surgical challenges and often unfavorable patient outcomes and high re-operation rate associated with the current treatment options for intracapsular femoral neck fractures.

This study will evaluate the re-operation rate for any reason of displaced and non-displaced femoral neck fractures treated with the CONQUEST FN Femoral Neck Fracture System at one year post-operation.

ELIGIBILITY:
Inclusion Criteria:

1. Must be 18 years of age or older
2. Must provide written informed consent
3. Willing to make all required study visits for one year post-operation
4. Subject has experienced a displaced or non-displaced intracapsular femoral neck fracture and is scheduled for repair using the CONQUEST FN Femoral Neck Fracture System.

Exclusion Criteria:

1. Subject with known sensitivity or allergies to stainless steel
2. Subject with fracture occurring more than 7 days prior to surgery
3. Subject has more than one fracture on the hip requiring surgery
4. Subject is considered obese by a Body Mass Index > 40 at the time of surgery
5. Therapy with another investigational agent within thirty 30 days of screening
6. Subject has emotional or neurological condition that precludes cooperation and compliance
7. Subject has undergone previous surgery on hip.
8. Subject has severe bow of the target hip or gross distortion of the femur.
9. Current systemic therapy with cytotoxic drugs
10. Subject has a physical condition that would preclude adequate implant support or impede healing (e.g. blood supply impairment, insufficient bone quality or quantity, or an active local or systemic infection).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-09-10 (Actual); Primary Completion 2020-02-11 (Actual); Study Completion 2020-02-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karlie Morgan, Study Chair — Smith & Nephew, Inc.
Locations (4):
- United States (4):
  - Orthopaedic Trauma Institute Navicent Health Medical Center, Macon, Georgia
  - Wake Forest School of Medicine, Winston-Salem, North Carolina
  - John Peter Smith Hospital, Fort Worth, Texas
  - UT Health Science Center San Antonio, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control Femoral Neck Fracture System
Started | 15
Completed | 3
Not Completed | 12
Not completed — Participant not able to return | 1
Not completed — Lost to Follow-up | 1
Not completed — Revision of the components of the study device | 2
Not completed — Sponsor terminated study | 6
Not completed — Death | 1
Not completed — Sponsor decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Control Femoral Neck Fracture System
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.9 (15.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White/caucasian | 14
  Race: Black/African American | 0
  Race: Asian | 0
  Race: Alaskan native/American indian | 0
  Race: Native Hawaiian/Other Pacific Islander | 0
  Race: Other | 1
Region of Enrollment [Number; unit: participants]
  United States | 15
Pre-injury Ambulatory Status [Count of Participants; unit: Participants]
  Unaided | 10
  Using a cane | 1
  Using a walker | 3
  Bed to chair | 1

OUTCOME MEASURES:

1. Primary Outcome: Reoperation Rate at One Year Post-operation
Description: Reoperation for any reason from time of implantation to one-year post operation
Time Frame: 1 year
Population: When study was terminated, only 3 participants completed their one year follow up visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Control Femoral Neck Fracture System
Number analyzed (Participants) | 3
Participants
  Reoperation | 2
  No Reoperation | 1

2. Secondary Outcome: Number of Participants With Intraoperative Complications
Description: Documentation of any complications related to the implantation of the device
Time Frame: 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Control Femoral Neck Fracture System
Number analyzed (Participants) | 15
Participants | 0

3. Secondary Outcome: Classification of Quality of Fracture Reduction
Description: Appropriate reduction was defined as the principal compressive trabeculae measuring >160° in the AP view and <5° of posterior angulation in the lateral view. Fractures were then classified as:
  * Grade I
  * Grade II
  * Grade III
  If reduction was acceptable in both views, it was classified as Grade I. Grade II was indicative of one plane of malreduction, and Grade III was indicative of malreduction in both radiographic views.
Time Frame: Operative, 6 weeks, 3 months, 6 months, and 1 year
Population: Number of Participants Analyzed indicates the data available for each given time frame as specified.
Measure: Count of Participants; unit: Participants
Arm/Group | Control Femoral Neck Fracture System
Number analyzed (Participants) | 15
Participants
  Operative: Grade I | 15
  Operative: Grade II | 0
  Operative: Grade III | 0
  6 weeks: number analyzed (Participants) | 12
  6 weeks: Grade I | 12
  6 weeks: Grade II | 0
  6 weeks: Grade III | 0
  3 months: number analyzed (Participants) | 10
  3 months: Grade I | 9
  3 months: Grade II | 0
  3 months: Grade III | 1
  6 months: number analyzed (Participants) | 4
  6 months: Grade I | 4
  6 months: Grade II | 0
  6 months: Grade III | 0
  1 year: number analyzed (Participants) | 3
  1 year: Grade I | 3
  1 year: Grade II | 0
  1 year: Grade III | 0

4. Secondary Outcome: Visual Analogue Scale (VAS) for Pain
Description: The Visual Analogue Scale was simply a line of fixed length, on which the subject marked their experience of pain with a single stroke of a pen. At each specified visit, the participant was asked to indicate their average level of pain from the operated hip over the prior 24 hours using a visual analog scale (VAS). The participant recorded their level of pain on a 100 millimeter visual analog scale with scores ranging from 0 to 100. The scale marked 'no pain' (score of 0) on the left side of the scale and 'severe pain' (score of 100) at the right end of the scale. The participant was instructed to place a vertical mark on the scale, using an ink pen.
  The Investigator, or designee, measured the distance (in millimeters) from the left end of the VAS scale to the vertical line drawn by the participant. This value was entered in the participant's Case Report Form (CRF) as a measure of the pain associated with the operated hip.
Time Frame: Pre-Operative, 6 Weeks, 3 Months, 6 Months, and 1 year
Population: Number Analyzed indicates available participant data for each time frame specified. Only 3 participants completed the 1 Year follow up visit when the study was terminated.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Femoral Neck Fracture System
Number analyzed (Participants) | 15
score on a scale
  Pre-Operative | 70.00 (28.06)
  6 Weeks: number analyzed (Participants) | 11
  6 Weeks | 32.30 (37.88)
  3 Months: number analyzed (Participants) | 10
  3 Months | 24.60 (29.79)
  6 Months: number analyzed (Participants) | 4
  6 Months | 12.50 (25.00)
  1 Year: number analyzed (Participants) | 3
  1 Year | 4.30 (1.53)

5. Secondary Outcome: Quality of Life - EQ-5D-5L
Description: The EuroQol Five Dimensions (EQ-5D-5L) Questionnaire descriptive system consists of 5 dimensions (mobility, self-care, usual activities, pain/discomfort and anxiety/depression), which are each assigned 5 levels:
  * 1= no problems
  * 2= slight problems
  * 3= moderate problems
  * 4= severe problems
  * 5= extreme problems
  The respondent is asked to indicate his/her health using the most appropriate statement in each of the 5 dimensions. This decision results in a 1-digit number expressing the level selected for that dimension. The digits for the five dimensions are combined in a 5-digit code describing the respondent's health state with scores ranging from -0.109 to 1 where higher scores indicate a better health state.
Time Frame: Pre-Operative, 6 Weeks, 3 Months, 6 Months, and 1 year
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Femoral Neck Fracture System
Number analyzed (Participants) | 15
score on a scale
  Pre-Operative | 0.3453 (0.3594)
  6 Weeks: number analyzed (Participants) | 11
  6 Weeks | 0.5164 (0.2612)
  3 Months: number analyzed (Participants) | 10
  3 Months | 0.6724 (0.2711)
  6 Months: number analyzed (Participants) | 4
  6 Months | 0.8938 (0.1366)
  1 Year: number analyzed (Participants) | 3
  1 Year | 0.8347 (0.1481)

6. Secondary Outcome: Timed Up and Go (TUG)
Description: The Timed Up and Go Test assesses mobility, balance, walking ability, and fall risk in adults by measuring time, in seconds, that it takes the individual to stand from a chair, walk a distance of 10 feet, walk back to the chair, and sit down. The subject will perform the test in their everyday footwear with their walking aid (cane, walker), if applicable. The site will follow the guidelines provided by the Centers for Disease Control and Prevention recording the results on the form provided by the Sponsor.
Time Frame: 6 Weeks, 3 Months, 6 Months, and 1 year
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Control Femoral Neck Fracture System
Number analyzed (Participants) | 8
seconds
  6 Weeks: number analyzed (Participants) | 7
  6 Weeks | 27.1 (17.09)
  3 Months | 31.4 (27.48)
  6 Months: number analyzed (Participants) | 4
  6 Months | 18.3 (10.53)
  1 Year: number analyzed (Participants) | 3
  1 Year | 14.3 (3.51)

7. Secondary Outcome: Active Straight Leg Raise (ASLR) Assessment: Evaluation Score
Description: The ASLR assessment provides information about the ability of load transfer and motor control strategies in the lumbo/pelvic/hip complex. ASLR will be performed with the subject in a relaxed supine position with legs straight and feet apart. Participants will be instructed to raise their operated leg 20cm above the examination table without bending the knee and without pelvic movement relative to the trunk. A score will be provided by the participant for the operated limb on a six-point Likert scale (0 = not difficult at all, 1 = minimally difficult; 2 = somewhat able to do, 3 = fairly difficult, 4 = very difficult, 5 = unable to do).
Time Frame: 6 Weeks, 3 Months, 6 Months, and 1 year
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Control Femoral Neck Fracture System
Number analyzed (Participants) | 12
Participants
  6 Weeks: 0- Not difficult at all | 5
  6 Weeks: 1- Minimally difficult | 2
  6 Weeks: 2- Somewhat able to do | 2
  6 Weeks: 3- Fairly difficult | 2
  6 Weeks: 4- Very difficult | 1
  6 Weeks: 5- Not able to do | 0
  3 Months: number analyzed (Participants) | 9
  3 Months: 0- Not difficult at all | 5
  3 Months: 1- Minimally difficult | 1
  3 Months: 2- Somewhat able to do | 1
  3 Months: 3- Fairly difficult | 1
  3 Months: 4- Very difficult | 1
  3 Months: 5- Not able to do | 0
  6 Months: number analyzed (Participants) | 4
  6 Months: 0- Not difficult at all | 3
  6 Months: 1- Minimally difficult | 1
  6 Months: 2- Somewhat able to do | 0
  6 Months: 3- Fairly difficult | 0
  6 Months: 4- Very difficult | 0
  6 Months: 5- Not able to do | 0
  1 Year: number analyzed (Participants) | 3
  1 Year: 0- Not difficult at all | 3
  1 Year: 1- Minimally difficult | 0
  1 Year: 2- Somewhat able to do | 0
  1 Year: 3- Fairly difficult | 0
  1 Year: 4- Very difficult | 0
  1 Year: 5- Not able to do | 0

8. Secondary Outcome: Number of Participants With Construct Failure
Description: Construct failure past typical femoral neck fracture healing period (past 6 months) indicated by reported device deficiencies.
Time Frame: 6 months post-operative
Population: Number Analyzed indicates available participant data for the time frame specified.
Measure: Count of Participants; unit: Participants
Arm/Group | Control Femoral Neck Fracture System
Number analyzed (Participants) | 4
Participants | 0

9. Secondary Outcome: Length of Hospital Stay
Description: Time spent in hospital measured by the number of days
Time Frame: During hospitalization
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Control Femoral Neck Fracture System
Number analyzed (Participants) | 15
days | 4.90 (1.83)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of surgery through the 1 year follow-up
Arm/Group | Control Femoral Neck Fracture System
All-Cause Mortality (participants affected / at risk) | 1/15
Serious Adverse Events (participants affected / at risk) | 5/15
Other Adverse Events (participants affected / at risk) | 3/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Femoral Neck Fracture System (N=15)
Screw fracture (Posterior, Proximal), Screw back out (Anterior, Proximal) (Product Issues) | 1 (1) — Device related
End stage Parkinson's Disease (Nervous system disorders) | 1 (1) — Not device related
St. Elevation Myocardial Infarction (Cardiac disorders) | 1 (1) — Not device related
Foot infection (Infections and infestations) | 1 (1) — Not device related
Non union (Product Issues) | 1 (1) — Device related
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Femoral Neck Fracture System (N=15)
Closed head injury (Injury, poisoning and procedural complications) | 1 (1) — Not device related
Ground level fall (Injury, poisoning and procedural complications) | 1 (1) — Not device related
Redness to right foot (Skin and subcutaneous tissue disorders) | 1 (1) — Not device related

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-30): https://cdn.clinicaltrials.gov/large-docs/35/NCT03721835/Prot_SAP_000.pdf